CLINICAL TRIAL: NCT00549978
Title: Phase IV, Safety and Pharmacokinetics of Probucol and Cilostazol When Coadministered in Healthy Subjects
Brief Title: Safety and Pharmacokinetics of Probucol and Cilostazol
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Korea Otsuka Pharmaceutical Co., Ltd. (Industry)
Collaborators: Otsuka Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 021-KOB-0702
Record Dates: First submitted 2007-10-25; First posted 2007-10-26 (Estimated); Last update posted 2022-03-04 (Actual); Status verified 2010-07

CONDITIONS: Healthy
Keywords: Safety and Pharmacokinetics in healthy subjects
MeSH Terms: interventions — Cilostazol; Probucol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Other): Two compartments with cross-over and parallel
  Interventions: Drug: Cilostazol
- 2 (Other): Two compartments with cross-over and parallel
  Interventions: Drug: Probucol

INTERVENTIONS:
Drug: Cilostazol — cilostazol, then cilostazol/probucol
  Arms: 1
Drug: Probucol — Probucol probucol/ cilostazol
  Arms: 2

SUMMARY:
to investigate the safety and pharmacokinetics, in healthy adult male subjects

DETAILED DESCRIPTION:
Safety and Pharmacokinetics of Probucol and Cilostazol when co-administered in Health Subjects

ELIGIBILITY:
Inclusion Criteria:

* Korean
* Gender: Male
* Age: Over 20 and Under 40years, at time of informed consent
* body weight: BMI over 19.0 and Under 25.0
* Subjects who meet the following criteria at the time of the screening examination
* Subjects who have given their written informed consent prior to participation in the study
* Subjects who are reliable and willing to make themselves available for the duration of the study and follow the study protocol

Exclusion Criteria:

* History or clinical evidence of significant respiratory, cardiovascular, renal, gastrointestinal, hepatic, endocrine, hematologic, neurologic, psychiatric, or other chronic disease, alcoholism, or drug abuse
* Present or previous significant drug allergy to any prescription or over the counter medication
* Blood collection exceeding 200ml within 4 weeks, 400ml within 12 weeks, or 1200ml within one year prior to scheduled study drug administration
* Body weight: under 50Kg

Ages: 20 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2007-10; Primary Completion 2008-05 (Actual); Study Completion 2008-08 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic parameters, Number of adverse events | during study follow-up period

SECONDARY OUTCOMES:
Physical exam, ECG, Vital signs and Laboratory tests, Drug interaction parameters | During study follow-up period

CONTACTS AND LOCATIONS:
Overall Officials: In-Jin Jang, PhD, Principal Investigator — Seoul National University Hospital
Locations (1):
- Clinical Trial Center, Seoul National University Hospital, Seoul, South Korea

REFERENCES:
- [Derived] Kim KP, Kim BH, Lim KS, Kim TE, Shin SG, Jang IJ, Yu KS. Potential interactions between cilostazol and probucol: a two-part, single-dose, open-label study in healthy Korean male volunteers. Clin Ther. 2009 Oct;31(10):2098-106. doi: 10.1016/j.clinthera.2009.10.005. PMID 19922880